CLINICAL TRIAL: NCT03647709
Title: Opioid-Free Accelerated Recovery Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: St. Elizabeth Medical Center, Utica, NY (Other)
Collaborators: Halyard Health (Industry)
Responsible Party: Principal Investigator, Dr Andrew B. Wickline, Orthopedic Surgeon, St. Elizabeth Medical Center, Utica, NY
Other Study IDs: qllS
Record Dates: First submitted 2018-08-09; First posted 2018-08-27 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Arthropathy of Knee Joint
MeSH Terms: interventions — Analgesics, Opioid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

INTERVENTIONS:
Other: opioids — dosage frequency and duration

SUMMARY:
To prove that total knee arthroplasty can be performed with little, if any need for opioids by using a combination of patient education, optimized pre-op and post-op pain and recovery protocols. The goal being opioid-free total knee arthroplasty.

DETAILED DESCRIPTION:
All study patients will receive a standardized protocol

* All surgical procedures performed by single surgeon using same implants, approach, pre-op and post-op optimization, and simplified pain protocol at a single hospital or surgery center
* Will attempt to minimize the number of anesthesiologists to further control variability in care

Methods:

1. Pre-op Optimization

   * All patients enroll in education program
   * All patients have optimized BMI, hemoglobin, albumin, glucose control-A1C, and blood pressure
2. Total Joint Procedure

   * Tourniquet-free cemented total knee arthroplasty is performed with intra-articular block
3. Data Collection

   * Electronic medical record chart review
   * Pre-op assessment and Post-op assessment (post anesthesia care unit (PACU), Phase II-prior to discharge
   * Phone calls after discharge
   * Follow-up assessment in surgeon's office
   * Swift path / KOOS JR surveys
4. Pain Management Regimen

   * pre-op physical therapy teaching
   * post-op multimodal pain regimen

ELIGIBILITY:
Inclusion Criteria:

* Surgeries to be performed at hospital
* Surgeries to be performed at surgery center
* Ability to read and understand English
* Primary care clearance for patients diagnosed with high blood pressure

Exclusion Criteria:

* Disease states, patient conditions to exclude:

Schizophrenia Bipolar Disease Dementia

* Known allergies to local anesthetics
* Previous burn to affected extremity
* BMI > 40
* Nonoptimized anemia
* Albumin less than 3.5
* A1C > 8.0

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A Partial and total knee arthroplasty Unilateral only
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Wickline, MD, Principal Investigator — St Elizabeth Medical Center
Locations (1):
- St Elizabeth Medical Center, Utica, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients to have total knee arthroplasty. All patients have optimized BMI, hemoglobin, albumin, glucose control-A1C and blood pressure. All patients enrolled in educational program. All patients have pre-op physical therapy teaching.
Groups:
- Total Knee Arthoplasty: All study patients received the same surgical procedure by the same surgeon, using same implants, approach, pre and post-optimization and a simplified pain protocol at a single hospital or surgery center.
  The number of opioid tablets taken by each patient was calculated from electronic medical record chart review, post anesthesia care unit, nursing care prior to discharge, phone calls after discharge and follow-up in surgeon's office.
Period: Overall Study
Arm/Group | Total Knee Arthoplasty
Started | 400
Completed | 386
Not Completed | 14
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Total Knee Arthroplasty: Number of patients that had total knee arthroplasty after meeting study inclusion criteria
Arm/Group | Total Knee Arthroplasty
Number analyzed (Participants) | 386
Age, Continuous [Median (Full Range); unit: years] | 69 [46 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226
  Male | 160
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m²] | 31.6 (5.2)
ASA [Number; unit: participants] — American Society of Anesthesiologists physical status classification system for assessing the fitness of patients before surgery. ASA I = normal healthy patient. ASA II = patient with mild systemic disease. ASA III = patient with severe systemic disease. ASA IV = patient with severe systemic disease that is a constant threat to life. Population: Number analyzed different from overall participants due to missing data from anesthesiologist record prior to surgery.
  participants
    I | 8
    II | 173
    III | 200
    IV | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Total Knee Replacement Performed Without Opioids Through 12 Weeks Postoperative
Description: Using a combination of patient education, optimized pre-operative and post-operative pain protocols and optimized recovery protocols
Time Frame: 12 weeks
Population: Number of patents that took no opioids after total knee arthroplasty 12 weeks post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Arthoplasty
Number analyzed (Participants) | 386
Participants | 73

2. Primary Outcome: Number of Patients With Total Knee Arthroplasty Performed With Opiate Drugs Through 12 Weeks Postoperative
Description: The total number of opioid tablets taken by patient after total knee arthroplasty performed through 12 weeks postoperative
Time Frame: 12 weeks
Population: Number of Participants Stratified by Total Quantity of Opioid Tablets Taken Post Total Knee Replacement
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Arthoplasty
Number analyzed (Participants) | 385
Participants
  no opioids | 72
  1-5 tablets | 159
  6-10 tablets | 101
  >10 tablets | 53

3. Secondary Outcome: Comparison of Change in Patient's Pain After Surgery At Various Time Intervals When Patient is at Rest and With Activity
Description: Pain level is measured by the Numerical Rating Scale (NRS) for pain utilizing minimum number 0 to maximum number 10 (0 represents no pain and 10 represents worst pain imaginable). The higher the number reported the worst the pain/outcome. This will be used to assess patient's level of pain relating to opioid use and recovery.
Time Frame: postoperative days 1,2,3,postoperative day 10-14, 3 weeks post surgery, 6 weeks post surgery and 12 weeks post surgery
Population: 386 patients analyzed through 6 weeks; 340 patients analyzed at 12 weeks only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Knee Arthoplasty
Number analyzed (Participants) | 386
score on a scale
  Postoperative Day 1 - Best with Rest | 1.0 (1.8)
  Postoperative Day 1 - Worst with Rest | 2.4 (2.3)
  Postoperative Day 1 - Best with Activity | 2.9 (2.2)
  Postoperative Day 1 - Worst with Activity | 4.6 (2.3)
  Postoperative Day 2 - Best at Rest | 1.8 (2.0)
  Postoperative Day 2 - Worst at Rest | 3.4 (2.3)
  Postoperative Day 2 - Best with Activity | 4.2 (2.0)
  Postoperative Day 2 - Worst with Activity | 5.9 (1.9)
  Postoperative Day 3 - Best at Rest | 1.0 (1.6)
  Postoperative Day 3 - Worst at Rest | 2.4 (2.1)
  Postoperative Day 3 - Best with Activity | 3.3 (2.1)
  Postoperative Day 3 - Worst with Activity | 5.0 (2.0)
  Postoperative Days 10-14 - Best at Rest | 0.5 (1.2)
  Postoperative Days 10-14 - Worst at Rest | 2.1 (2.0)
  Postoperative Days 10-14 - Best with Activity | 2.0 (1.9)
  Postoperative Days 10-14 Worst with Activity | 4.0 (2.1)
  Postoperative Week 3 - Best at Rest | 0.3 (0.8)
  Postoperative Week 3 - Worst at Rest | 1.5 (1.9)
  Postoperative Week 3- Best with Activity | 1.3 (1.6)
  Postoperative Week 3 - Worst with Activity | 3.1 (2.1)
  Postoperative Week 6 - Best at Rest | 0.1 (0.6)
  Postoperative Week 6 - Worst at Rest | 0.7 (1.5)
  Postoperative Week 6 - Best with Activity | 0.5 (1.2)
  Postoperative Week 6 - Worst with Activity | 1.9 (2.0)
  Postoperative Week 12 - Best at Rest: number analyzed (Participants) | 340
  Postoperative Week 12 - Best at Rest | 0.0 (0.2)
  Postoperative Week 12 - Worst at Rest: number analyzed (Participants) | 340
  Postoperative Week 12 - Worst at Rest | 0.2 (0.7)
  Postoperative Week 12 - Best with Activity: number analyzed (Participants) | 340
  Postoperative Week 12 - Best with Activity | 0.0 (0.3)
  Postoperative Week 12 - Worst with Activity: number analyzed (Participants) | 340
  Postoperative Week 12 - Worst with Activity | 0.5 (1.2)
Statistical Analysis 1: Comparison: Total Knee Arthoplasty; Comparison of change in patient's reported pain with rest or during activity at various time intervals. Patients reported best and worst pain scores at rest and during activity; Test type: Other; mean score = 1.0, 95% CI 2-sided [0.9 to 1.2] — Represents patients pain score post operative day 1 best with rest
Statistical Analysis 2: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 2.4, 95% CI 2-sided [2.2 to 2.6] — Represents patients reported pain score post operative day 1 worst at rest
Statistical Analysis 3: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 2.9, 95% CI 2-sided [2.7 to 3.1] — Represents patients reported pain score post operative day 1 best with activity
Statistical Analysis 4: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 4.6, 95% CI 2-sided [4.4 to 4.8] — Represents patients reported pain score post operative day 1 worst with activity
Statistical Analysis 5: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 1.8, 95% CI 2-sided [1.6 to 2.0] — Represents patients reported pain score post operative day 2 best at rest
Statistical Analysis 6: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 3.4, 95% CI 2-sided [3.2 to 3.6] — Represents patients reported pain score post operative day 2 worst at rest
Statistical Analysis 7: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 4.2, 95% CI 2-sided [4.0 to 4.4] — Represents patients reported pain score post operative day 2 best with activity
Statistical Analysis 8: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 5.9, 95% CI 2-sided [5.7 to 6.1] — Represents patients reported pain score post operative day 2 worst with activity
Statistical Analysis 9: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 1.0, 95% CI 2-sided [0.8 to 1.2] — Represents patients reported pain score post operative day 3 best at rest
Statistical Analysis 10: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 2.4, 95% CI 2-sided [2.2 to 2.6] — Represents patients reported pain score post operative day 3 worst at rest
Statistical Analysis 11: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 3.3, 95% CI 2-sided [3.1 to 3.5] — Represents patients reported pain score post operative day 3 best with activity
Statistical Analysis 12: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 5.0, 95% CI 2-sided [4.8 to 5.2] — Represents patients reported pain score post operative day 3 worst with activity
Statistical Analysis 13: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.5, 95% CI 2-sided [0.4 to 0.7] — Represents patients reported pain score post operative days 10-14 best at rest
Statistical Analysis 14: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 2.1, 95% CI 2-sided [1.9 to 2.3] — Represents patients reported pain score post operative days 10-14 worst at rest
Statistical Analysis 15: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 2.0, 95% CI 2-sided [1.8 to 2.2] — Represents patients reported pain score post operative days 10-14 best with activity
Statistical Analysis 16: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 4.0, 95% CI 2-sided [3.8 to 4.2] — Represents patients reported pain score post operative days 10-14 worst with activity
Statistical Analysis 17: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.3, 95% CI 2-sided [0.2 to 0.4] — Represents patients reported pain score post operative week 3 best at rest
Statistical Analysis 18: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 1.5, 95% CI 2-sided [1.3 to 1.7] — Represents patients reported pain score post operative week 3 worst at rest
Statistical Analysis 19: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 1.3, 95% CI 2-sided [1.2 to 1.5] — Represents patients reported pain score post operative week 3 best with activity
Statistical Analysis 20: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 3.1, 95% CI 2-sided [2.9 to 3.3] — Represents patients reported pain score post operative week 3 worst with activity
Statistical Analysis 21: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.1, 95% CI 2-sided [0.0 to 0.2] — Represents patients reported pain score post operative week 6 best at rest
Statistical Analysis 22: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.7, 95% CI 2-sided [0.5 to 0.8] — Represents patients reported pain score post operative week 6 worst at rest
Statistical Analysis 23: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.5, 95% CI 2-sided [0.4 to 0.6] — Represents patients reported pain score post operative week 6 best with activity
Statistical Analysis 24: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 1.9, 95% CI 2-sided [1.7 to 2.0] — Represents patients reported pain score post operative week 6 worst with activity
Statistical Analysis 25: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.0, 95% CI 2-sided [-0.0 to 0.0] — Represents patients reported pain score post operative week 12 best at rest
Statistical Analysis 26: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.2, 95% CI 2-sided [0.1 to 0.2] — Represents patients reported pain score post operative week 12 worst at rest
Statistical Analysis 27: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.0, 95% CI 2-sided [-0.0 to 0.1] — Represents patients reported pain score post operative week 12 best with activity
Statistical Analysis 28: Comparison: Total Knee Arthoplasty; [analysis description as in outcome 3, analysis 1]; Test type: Other; mean score = 0.5, 95% CI 2-sided [0.4 to 0.7] — Represents patients reported pain score post operative week 12 worst with activity

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score Short Form (KOOS JR)
Description: The Knee Injury and Osteoarthritis Outcome Score Short Form (KOOS JR) is a survey that is an assessment and questionnaire that rates a patients joint pain, stiffness and function in daily living. Patients answer questions about joint stiffness, pain and daily activities using the following scoring values: 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme. The values for all questions are added up to get a raw score that ranges from a minimum of 0 to a maximum of 28. This raw score is converted to an interval score using a provided table. The interval score ranges from a minimum of 0 to a maximum of 100 where 0 = total knee disability and 100 = perfect knee health. The higher the score on scale from 0 to 100 the better the outcome.
Time Frame: Baseline (preoperative); 6 weeks post surgery; 12 weeks post surgery
Population: 311 patients reported KOOS JR scores at baseline which was prior to surgery. At 6 weeks 379 patients reported scores. At 12 weeks 341 patients reported scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Knee Arthoplasty
Number analyzed (Participants) | 379
score on a scale
  Baseline prior to surgery: number analyzed (Participants) | 311
  Baseline prior to surgery | 53.1 (11.9)
  Postoperative 6 Week | 71.8 (11.8)
  Postoperative 12 Week: number analyzed (Participants) | 341
  Postoperative 12 Week | 90.0 (8.2)

5. Secondary Outcome: Number of Participants Using Swift Path Educational Tool as Outpatients for Total Joint Replacement
Description: Swift path is an Educational tool (diary) for patients undergoing total joint replacement, that patients follow from the initial booking of surgery through their recovery. It guides patients through potential risks involved with joint surgery, through a multimodal pain management protocol for pain prevention and through recovery.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Total Knee Arthoplasty
Number analyzed (Participants) | 386
Participants | 386

6. Secondary Outcome: Number of Patients That Adhered to Exercise Protocol After Having Total Knee Arthroplasty - Postop Days 10-14
Description: Exercise protocol for patients after total knee replacement where the patient performs a series of exercises every hour to help prevent blood clots and achieve appropriate range of motion goals.
Time Frame: Postop Days10-14
Population: Physical therapy adherence for patients not taking opioids and taking opioids at 10-14 day follow-up visit
Measure: Count of Participants; unit: Participants
Groups:
- No Opiates and Physical Therapy Adherence: Physical therapy adherence and non adherence for follow-up visits (1) post surgery days 10-14; (2) 3 weeks post surgery; (3) 6 weeks post surgery; (4) 12 weeks post surgery
- Opiates and Physical Therapy Adherence: physical therapy adherence and non-adherence Post surgery Days 10-14, week 3 post surgery, 6 week post surgery and 12 week post surgery
Arm/Group | No Opiates and Physical Therapy Adherence | Opiates and Physical Therapy Adherence
Number analyzed (Participants) | 269 | 117
Participants
  PT Adherence | 193 | 64
  PT Non-adherence | 76 | 53
Statistical Analysis 1: Comparison: No Opiates and Physical Therapy Adherence vs Opiates and Physical Therapy Adherence; Test type: Other; p = 0.0015, Fisher Exact

7. Secondary Outcome: Number of Patients That Adhered to Exercise Protocol After Having Total Knee Arthroplasty - Postop Week 3
Description: as for outcome 6
Time Frame: postoperative 3 weeks
Population: Physical therapy adherence for patients not taking opioids and taking opioids at 3 week follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | No Opiates and Physical Therapy Adherence | Opiates and Physical Therapy Adherence
Number analyzed (Participants) | 349 | 35
Participants
  PT Adherence | 290 | 28
  PT Non-adherence | 59 | 7
Statistical Analysis 1: Comparison: No Opiates and Physical Therapy Adherence vs Opiates and Physical Therapy Adherence; Test type: Other; p = .6398, Fisher Exact

8. Secondary Outcome: Number of Patients That Adhered to Exercise Protocol After Having Total Knee Arthroplasty - Postop Week 6
Description: as for outcome 6
Time Frame: Postoperative 6 weeks
Population: Physical therapy adherence for patients not taking opioids and taking opioids at 6 week follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | No Opiates and Physical Therapy Adherence | Opiates and Physical Therapy Adherence
Number analyzed (Participants) | 373 | 12
Participants
  PT Adherence | 361 | 10
  PT Non-adherence | 12 | 2
Statistical Analysis 1: Comparison: No Opiates and Physical Therapy Adherence vs Opiates and Physical Therapy Adherence; Test type: Other; p = .0658, Fisher Exact

9. Secondary Outcome: Number of Patients That Adhered to Exercise Protocol After Having Total Knee Arthroplasty - Post Week 12
Description: as for outcome 6
Time Frame: Postoperative 12 weeks
Population: Physical therapy adherence for patients not taking opioids and taking opioids at 12 week follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | No Opiates and Physical Therapy Adherence | Opiates and Physical Therapy Adherence
Number analyzed (Participants) | 335 | 2
Participants
  PT Adherence | 297 | 2
  PT Non-adherence | 38 | 0
Statistical Analysis 1: Comparison: No Opiates and Physical Therapy Adherence vs Opiates and Physical Therapy Adherence; Test type: Other; p = 1.0000, Fisher Exact

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were events that occurred from day of surgery through 12 week post-surgery.
Arm/Group | Total Knee Arthoplasty
All-Cause Mortality (participants affected / at risk) | 0/386
Serious Adverse Events (participants affected / at risk) | 4/386
Other Adverse Events (participants affected / at risk) | 33/386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Knee Arthoplasty (N=386)
infection (Infections and infestations) | 1 (1) — patient had post surgery incision and drainage of acute total knee arthroplasty infection week 4 and placed on antibiotics.
right quadricep repair (Musculoskeletal and connective tissue disorders) | 1 (1) — patient experienced right quadriceps repair which was torn during formal physical therapy post surgery week 8
bowel obstruction (Gastrointestinal disorders) | 1 (1) — not related to surgery Patient had a history of bowel obstruction
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — unrelated to surgery occurred during patient rehab stay
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Knee Arthoplasty (N=386)
bleeding (Skin and subcutaneous tissue disorders) | 2 (2) — bleeding from suture site which required a pressure bandage to control further bleeding
fall (Social circumstances) | 14 (14) — patient reported a fall (none resulted in an intervention or injuries)
motor weakness (Surgical and medical procedures) | 8 (8) — motor weakness due to adductor canal anesthesia/numbness
paresthesia (Nervous system disorders) | 1 (1) — persistent patient had history of multiple sclerosis prior to surgery
uncontrolled pain (Surgical and medical procedures) | 4 (4) — persistent pain post surgery which included nerve pain and burning
early pain ball catheter removal by patient (Surgical and medical procedures) | 9 (9) — patients removed pain ball prior to completion due to leakage or mechanical problem
inadvertent pain ball catheter removal (Surgical and medical procedures) | 3 (3) — patient removed pain ball or disconnected pain ball by mistake
persistent numbness (Nervous system disorders) | 2 (2) — patient experiencing numbness to touch
manipulation of knee joint (Musculoskeletal and connective tissue disorders) | 9 (9) — patients required manipulation of knee joint due to poor range of motion of knee post surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03647709/Prot_000.pdf